CLINICAL TRIAL: NCT02067871
Title: Neuromuscular Electrical Stimulation and Low-level Laser: Combined Use for the Treatment of Knee Osteoarthritis in Elderly
Brief Title: Treatment of Knee Osteoarthritis: Neuromuscular Electrical Stimulation and Low-level Laser.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Aurélio Vaz, PhD (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS - 20160
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Knee Osteoarthritis
Keywords: neuromuscular electrical stimulation; low-level laser therapy; knee osteoarthritis; muscle architecture; functionality; neuromuscular parameters
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Laser Therapy; Low-Level Light Therapy; Phototherapy; Electric Stimulation; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electrical stimulation (Experimental): * 18-32 min of pulsed current.
  * stimulation frequency of 80Hz (hertz).
  * pulse duration of 200μs (microseconds).
  * stimulation intensity fixed near to maximal tolerated.
  Interventions: Other: Electrical Stimulation
- Laser Therapy (Experimental): * λ = 810 nm (nanometers)
  * continuous wave
  * 200 mW (milliwatts) output power
  * low-level laser therapy dose of 4-6J (Joules) per point
  * six points at the knee joint
  Interventions: Other: Laser Therapy
- Combined Treatment (Experimental): Electrical Stimulation:
  * 18-32 min of pulsed current,
  * stimulation frequency of 80Hz (hertz).
  * pulse duration of 200μs (microseconds).
  * stimulation intensity fixed near to maximal tolerated.
  and
  Laser Therapy:
  * λ = 810 nm (nanometers)
  * continuous wave
  * 200 mW (milliwatts) output power
  * low-level laser therapy dose of 4-6J (Joules) per point.
  * six points at the knee joint.
  Interventions: Other: Laser Therapy; Other: Electrical Stimulation

INTERVENTIONS:
Other: Laser Therapy — Low-level laser therapy was administered twice a week with a minimum of 48h between sessions over a period of eight weeks.
  Other Names: Low-Level Laser Therapy; Lasertherapy; Light therapy; Phototherapy
  Arms: Combined Treatment; Laser Therapy
Other: Electrical Stimulation — Neuromuscular electrical stimulation was administered twice a week with a minimum of 48h between sessions over a period of eight weeks and with progressive intensity and volume.
  Other Names: electrotherapy; electrical stimulation therapy; neuromuscular electrical stimulation
  Arms: Combined Treatment; Electrical stimulation

SUMMARY:
* The purpose of this study is to determine the effects of low-level laser therapy in combination with neuromuscular electrical stimulation on neuromuscular (muscular strength and morphology) and functional parameters (pain and functional tests) in elderly with knee osteoarthritis.
* The hypothesis is that the association of low-level laser therapy with neuromuscular electrical stimulation could reduce joint pain associated with the inflammation and consequently potentiates the effects of electrical stimulation on the muscular system.

DETAILED DESCRIPTION:
* Participants was randomized into one of three intervention groups (intervention period = 8 weeks after a 4 weeks control period in all groups).
* Electrical stimulation group (18-32 min of pulsed current, stimulation frequency of 80Hz (Hertz), pulse duration of 200μs and stimulation intensity fixed near to maximal tolerated),
* Laser group (low-level laser therapy dose of 4-6J (Joules) per point, six points at the knee joint)
* Combined group (electrical stimulation and low-level laser therapy).

ELIGIBILITY:
Inclusion Criteria:

* elderly.
* symptomatic knee osteoarthritis.
* radiographic diagnostic of Grade 2 or 3 knee osteoarthritis.

Exclusion Criteria:

* a body mass index higher than 40 Kg/m2.
* a diagnosis of hip, ankle, or toe osteoarthritis.
* the use of crutches for locomotion.
* participation in a strength-training programme or physiotherapy treatment for knee osteoarthritis in the past six months.
* neurological or cognitive disorders.
* rheumatoid arthritis.
* electronic implants.
* previous or upcoming surgery (within three months).
* any cardiorespiratory, neuromuscular, or metabolic disease that could represent an absolute contraindication or a contraindication to the performance of maximum strength tests.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Torque change | Torque was measured 3 times during the study: baseline (week -4), before intervention (week 0) and post intervention (week 9).
  Torque is an expression of the muscular strength and was assessed by dynamometry.

SECONDARY OUTCOMES:
Muscular architecture change | Architecture was measured 3 times during the study: baseline (week -4), before intervention (week 0) and post intervention (week 9).
  Muscular architecture (muscle thickness, pennation angle and fascicle length) were assessed by ultrasonography.

OTHER OUTCOMES:
Functional Performance change | Functional performace was measured 3 times during the study: baseline (week -4), before intervention (week 0) and post intervention (week 9).
  Functional performance was assessed using the six-minute walk test and the Timed Up and Go test.
Pain Change | Pain was measured 3 times during the study: baseline (week -4), before intervention (week 0) and post intervention (week 9).
  Pain was assessed by questionnaire
Muscular electrical activation change | Muscular electrical activation was measured 3 times during the study: baseline (week -4), before intervention (week 0) and post intervention (week 9)
  Electrical activation was assessed by electromyography (EMG).

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil